CLINICAL TRIAL: NCT05058157
Title: Ketone Plasma Kinetics After Oral Intake of Different Ketogenic Formulae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1803NR
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Healthy Men and Women

STUDY DESIGN:
Intervention Model Description: Each testing cycle design will be either a complete or partial cross-over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ketone Precursor Formula 1 (Active Comparator): Formula 1 (in each cycle, up to 4 formula will be tested) Ketone precursors formula (powder to reconstitute in drinking water, or in a ready-to-drink format).
  Interventions: Dietary Supplement: different ketogenic formulae
- Ketone Precursor Formula 2 (Active Comparator): Ketone precursors formula (powder to Reconstitute in drinking water, or in a ready-to-drink format).
  Interventions: Dietary Supplement: different ketogenic formulae
- Ketone Precursor Formula 3 (Active Comparator): Ketone precursors formula (powder to Reconstitute in drinking water, or in a ready-to-drink format)
  Interventions: Dietary Supplement: different ketogenic formulae
- Ketone Precursor Formula 4 (Active Comparator): Ketone precursors formula (powder to Reconstitute in drinking water, or in a ready-to-drink format), or placebo
  Interventions: Dietary Supplement: different ketogenic formulae

INTERVENTIONS:
Dietary Supplement: different ketogenic formulae — The research product may be in a form of powder to reconstitute or in a ready-to-drink format.

SUMMARY:
This research project aims at evaluating the effect of various ketone precursors and their formulations on blood ketone level after oral intake. Evaluation of the GI tolerability of the various formula will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, based on the screening visit and medical history,
* BMI in the normal and overweight range 18.5 ≤ BMI ≤ 27;
* Able to understand and sign informed consent form.

Exclusion Criteria:

* Any medication possibly impacting the postprandial glucose and insulin response (based on anamnesis),
* Any medication impacting dietary fat absorption and metabolism,
* Pregnancy (on anamnesis) and/or lactation,
* Known food allergy and food intolerance,
* Individuals undergoing either dietary or exercise mediated weight loss program prescribed by a health care professional,
* Individuals under ketogenic diets, or taking regular ketones products,
* Alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of bier,
* Having given blood within the last month, or willing to make a blood donation until one month following the end of the study,
* Family or hierarchical relationships with Clinical Innovation Lab at Nestlé Research, Lausanne, Switzerland,
* Volunteer who cannot be expected to comply with the protocol,
* Smokers unable to stop for the day of the visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Ketone Plasma Kinetics After Oral Intake of Different Ketogenic Formulae | 0 (baseline) to 4 hours after products consumption
  Incremental area under the curve of total blood ketones

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Sun, Principal Investigator — Société des Produits Nestlé (SPN)
Locations (1):
- Nestlé Clinical Innovation Lab, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided